CLINICAL TRIAL: NCT03340948
Title: The Mindfulness Intervention as Myocardial Infarction Rehabilitation Additive (MIMIRA) Study
Acronym: MIMIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Oskar Lundgren, PhD Candidate, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013/17/31
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Disease; Depressive Symptoms
Keywords: Mindfulness Based Stress Reduction; Depressive symptoms; Coronary Artery Disease; Mastery
MeSH Terms: conditions — Coronary Artery Disease; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Pilot and feasibility study of one cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBSR participation (Experimental): Participation in the 8 week Mindfulness Based Stress Reduction (MBSR) course.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — An 8-week course in mindfulness meditation, yoga training and weekly group support in the form of weekly 2,5 hour meetings at the hospital.

SUMMARY:
The Mindfulness Intervention as Myocardial Infarction Rehabilitation Additive (MIMIRA) study aimed at studying the feasibility and acceptability of Mindfulness Based Stress Reduction - an 8 week course in meditation and yoga - in patients with a recent coronary artery event and elevated depressive symptoms. To address these questions patients with elevated scores on a depression scale were invited to participate in MBSR, and there evaluation of the course as well as a panel of psychological risk factors and resources was measured.

DETAILED DESCRIPTION:
Depressive symptomatology in patients with coronary artery disease (CAD) has prognostic importance. Yet, psychological interventions in clinical practice are scarce. Here, we explored the feasibility and acceptability of mindfulness-based stress reduction (MBSR) in patients with depressive symptoms after a recent coronary event. A second aim was to investigate psychological risk factors and resources among participants.

To address the research questions, depressive symptoms were first measured in a reference population, at 1 and 12 months after a coronary event (myocardial infarction or unstable angina pectoris), and a cut-off for elevated depressive symptoms were obtained from the median in this group. Thereafter, similar CAD patients with elevated depressive symptoms (above median in the reference group), from the same outpatient clinic, were consecutively invited to an 8-week MBSR program. Serious physical or psychiatric illness that would be an obstacle to participation were exclusion criteria.

Patients who completed the MBSR-course were asked to evaluate its various facets, and completion rate and attendance were feasibility outcomes. Psychological variables were measured before, after the course as well as 12 months later.

ELIGIBILITY:
Inclusion Criteria:

1. Recent (within 12 month) first time coronary artery event; defined as a diagnosis of myocardial infarction or unstable angina pectoris addressed with either percutaneous coronary intervention (PCI) or coronary artery by-pass graft surgery (CABG).
2. Depressive symptoms above a score of 8 on the questionnaire centre for epidemiological studies depression scale (CES-D).
3. Interest for participation in MBSR.

Exclusion Criteria:

1. Major depression or other serious psychiatric illness (such as psychosis or ongoing life crisis).
2. Severe comorbidities, such as cancer, severe cognitive impairment and alcohol or drug abuse.
3. Practical hindrances for participation in MBSR.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01-31 (Actual); Primary Completion 2014-11-18 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility | Immediately after the 8-week intervention.
  Patient evaluation questionnaire

SECONDARY OUTCOMES:
Depressive Symptoms | Before, immediately after and 12 months post intervention.
  Centre for Epidemiological Studies Scale Depression (CES-D) questionnaire (Radloff)
Anxiety | Before, immediately after and 12 months post intervention.
  Generalized Anxiety Disorder Scale - 7 (GAD-7) questionnaire (Spitzer)
Mindfulness | Before, immediately after and 12 months post intervention.
  Five Facets of Mindfulness Questionnaire (FFMQ) (Baer)
Acceptance | Before, immediately after and 12 months post intervention.
  Acceptance and Action Questionnaire II (AAQII) (Block)
Mastery | Before, immediately after and 12 months post intervention.
  Mastery questionnaire (Pearlin & Shooler)
Self-esteem | Before, immediately after and 12 months post intervention.
  Self-esteem questionnaire (Rosenberg)
Patients experiences of mindfulness training | Continuously during the 8 week course.
  Written journal entries (linguistic content)

CONTACTS AND LOCATIONS:
Overall Officials: Lena LJ Jonasson, M.D. Ph.D., Principal Investigator — Division of Cardiovascular Medicine, Department of Medical and Health Sciences, Linköping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available on reasonable request.

REFERENCES:
- [Derived] Lundgren O, Garvin P, Nilsson L, Tornerefelt V, Andersson G, Kristenson M, Jonasson L. Mindfulness-Based Stress Reduction for Coronary Artery Disease Patients: Potential Improvements in Mastery and Depressive Symptoms. J Clin Psychol Med Settings. 2022 Sep;29(3):489-497. doi: 10.1007/s10880-021-09822-z. Epub 2021 Sep 28. PMID 34585329
- [Derived] Lundgren O, Garvin P, Kristenson M, Jonasson L, Thylen I. A journey through chaos and calmness: experiences of mindfulness training in patients with depressive symptoms after a recent coronary event - a qualitative diary content analysis. BMC Psychol. 2018 Sep 13;6(1):46. doi: 10.1186/s40359-018-0252-1. PMID 30213276